CLINICAL TRIAL: NCT02309060
Title: Narrative Intervention to Disseminate ACT for Depression in Primary Care
Brief Title: Storytelling Video Intervention for Depressed Primary Care Patients - Open Trial
Acronym: sTVi-Open
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Uebelacker, Co-PI, Butler Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sTVi-1; R34MH103568 (NIH)
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Major Depressive Disorder
Keywords: narrative communication; depression; primary care; treatment development
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Storytelling Video Intervention (sTVi) (Experimental): We will develop a series of 4 videos, each episode approximately 30 minutes long, which will illustrate the key principles of Acceptance and Commitment Therapy.
  We will add a short, non-narrative, epilogue at the end of each of the 4 episodes that summarizes key messages and provides information on identifying signs of depression and suggestions for efficacious treatments.
  In addition, we will develop an accompanying "personal journal" for participants that includes a brief self-help guide which encourages participants to write about what they learned in the videos and how they will take similar steps in their own lives to cope with depression.
  Interventions: Behavioral: Storytelling Video Intervention (sTVi)

INTERVENTIONS:
Behavioral: Storytelling Video Intervention (sTVi) — Narrative communication, video-based intervention for depressed primary care patients.

SUMMARY:
The overall aim of this program of research is to develop a collaborative narrative intervention for patients with depression being treated in primary care.

The purpose of the proposed project is to establish the feasibility, acceptability, and preliminary effects of our newly developed narrative intervention on depression.

To achieve the specific aims, the investigators will conduct an open trial to further develop and refine the intervention (n = 10).

DETAILED DESCRIPTION:
The public health impact of existing treatments for major depression is limited by our ability to disseminate those treatments. There is a particular need to find innovative ways to disseminate key principles of empirically supported psychotherapy in primary care settings. Narrative communication is an alternative way to disseminate psychotherapy behavior change principles. Narrative communication refers to "storytelling" -real people talking about their struggles and successful ways of coping. An advantage of narrative communication is that it can be easily distributed (by video) and may reach people who do not have access to other technologies or who experience barriers to traditional psychotherapy. We propose that key principles of a type of cognitive-behavioral therapy (Acceptance and Commitment Therapy, or ACT) can be readily disseminated through a video storytelling intervention. ACT is an empirically supported therapy for depression. Together with a video production firm with a record of working in healthcare and developing documentary-style videos, we will produce a storytelling video intervention (sTVi).

Our aim is to conduct a small open trial (n = 10) of antidepressant medication treatment as usual + sTVi. Assessments will occur at baseline and 4 weeks (post-treatment). We will examine the feasibility and acceptability of sTVi (e.g., uptake and completion of sTVi, engagement with videos, and understanding of key ACT principles) and of this research design. We will examine treatment effects (within relevant confidence intervals) on outcomes (e.g., depression severity). We will examine change in potential mechanisms, i.e., ACT-consistent coping strategies derived from key ACT principles.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-5 criteria for current or lifetime major depressive disorder.
2. No Lifetime diagnosis of bipolar disorder, schizophrenia, or chronic psychotic condition.
3. No current hazardous illicit drug or alcohol use.
4. No suicidal ideation or behavior requiring immediate attention.
5. Depression symptom severity: a Quick Inventory of Depressive Symptoms (QIDS) score >11.
6. Taking an antidepressant medication for at least 6 weeks; prescribed by their primary care provider.
7. Not in psychotherapy during the study period.
8. Have a PCP at our enrollment site.
9. If pregnant, less than 24 weeks gestation.
10. English speaking.
11. Aged 18 or older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire-8 (CSQ-8) | 4 weeks

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology-Clinician Rating (QIDS-C) | 4 weeks
Acceptance and Action Questionnaire-II (AAQ-II) | 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital/Brown University; Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital/Brown University
Locations (2):
- United States (2):
  - Family Care Center of Memorial Hospital, Pawtucket, Rhode Island
  - Butler Hospital, Providence, Rhode Island

REFERENCES:
- [Result] Gaudiano BA, Davis CH, Miller IW, Uebelacker LA. Development of a Storytelling Video Self-Help Intervention Based on Acceptance and Commitment Therapy for Major Depression: Open Trial Results. Behav Modif. 2019 Jan;43(1):56-81. doi: 10.1177/0145445517738932. Epub 2017 Nov 1. PMID 29090593